CLINICAL TRIAL: NCT06929559
Title: Muscular Synergies and Behavioral Adaptations of Gait in Pain Anticipation (SYAMAPP)
Acronym: SYAMAPP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universite de Picardie Jules Verne (Other)
Responsible Party: Principal Investigator, Jennifer Burgos Tirado, Researcher - Ph.D student, Universite de Picardie Jules Verne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB00012476-2025-26-03-393
Record Dates: First submitted 2025-03-27; First posted 2025-04-16 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Nocebo Effect; Pain Anticipation
Keywords: Nocebo effect; Pain anticipation; Pain expectation; Motricity; Gait; Walking; Healthy; Muscle synergies
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are not aware that a cream applied to them (neutral cream) does not produce any pain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nocebo Conditioning Group (Experimental): Participants in this arm will receive the neutral cream with instructions suggesting it may cause pain.
  Interventions: Other: Pain expectation conditioning; Other: Intervention: Gait
- Control Group (Placebo Comparator): Participants receive application of identical neutral cream with verbal and behavioral suggestions that it may cause localized pain, creating a nocebo effect through expectation manipulation.
  Interventions: Other: Comparator (Control Group); Other: Intervention: Gait

INTERVENTIONS:
Other: Pain expectation conditioning — Participants receive application of a neutral cream (MEDICAFARM) with verbal and behavioral suggestions that it may cause localized pain. Researchers wear gloves during application and emphasize potential discomfort, stating effects may intensify with movement.
  Arms: Nocebo Conditioning Group
Other: Comparator (Control Group) — Participants receive identical application of the neutral cream but are informed it is inert and harmless. Researchers apply the cream without gloves and provide neutral instructions.
  Arms: Control Group
Other: Intervention: Gait — Participants undergo assessment procedures including:
  * Pre- and post-application gait analysis (GAITRite mat, Zebris treadmill)
  * Physiological monitoring (EMG, HRV, EDA)
  * Identical questionnaires (BPI, TSK, FACS, PCS, VAS)

SUMMARY:
The purpose of this study is to determine whether the anticipation of pain influences gait control and psychophysiological responses in healthy individuals. Participants will receive a neutral cream described either as potentially painful (experimental group) or inert (control group), and their behavioral and physiological adaptations will be measured during walking tasks.

DETAILED DESCRIPTION:
Pain anticipation can significantly alter motor behavior and physiological responses, even in the absence of actual pain. While previous research has established that conditioned expectations can modify gait patterns, muscle activation, and autonomic responses, the specific locomotor adaptations triggered by pain anticipation in healthy individuals remain insufficiently understood. This study examines how manipulating expectations about a neutral cream influences gait control and psychophysiological markers during walking tasks.

Participants will be recruited through university announcements including posters and emails, with eligibility determined via an online screening questionnaire and verbal confirmation the day of the experience. Healthy adults aged 18-35 who meet the inclusion criteria will participate in a single 90-minute experimental session. Random assignment will place participants into either an experimental group, where they receive the neutral cream with verbal suggestions that it may cause localized pain, or a control group that receives identical application with neutral instructions.

The experimental protocol consists of two primary walking assessments conducted both before and after cream application. First, participants perform free walking trials on a GAITRite mat to measure baseline spatiotemporal parameters including walking speed, cadence, and step length at a comfortable speed until completion of 30 gait cycles. Second, treadmill walking and running trials using a Zebris system evaluate gait transitions through incremental speed changes from 0.5 m/s to 4.1 m/s in increments of 0.4 m/s with 10 second familiarisation time in-between measurements. Both walking tasks are recorded using GoPro cameras to subsequent analysis of changes in joint amplitudes. Throughout these tasks, physiological monitoring captures muscle activity via surface EMG, cardiac responses through ECG and heart rate variability measurements, and electrodermal activity as an indicator of autonomic arousal.

Following the first movement assessments and before the application of the cream, participants complete standardized questionnaires evaluating pain perception using the Brief Pain Inventory and visual analog scales (VAS), fear of movement through the Tampa Scale of Kinesiophobia and Fear-Avoidance Components Scale, and pain catastrophizing via the Pain Catastrophizing Scale.

The cream is applied at the level of the knee, between the two lateral epicondyles of the femur with a 4 cm width, and another VAS is filled in after application. The walking tasks are repeated, measuring the same physiological signs and three more VAS's are administered: one during the treadmill walking task, at the end of the 1.3 m/s speed recording, another during the free walking task, after half of the completed gait cycles, and a final one at the end of the protocol.

The primary outcome measure focuses on changes in the walk ratio, calculated as step length divided by cadence, while secondary outcomes examine alterations in kinematic patterns, muscle activation strategies, and autonomic nervous system responses.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-35 years
* Healthy participant with no self-reported diagnosed neurological, musculoskeletal, or cardiovascular disorders
* Body Mass Index (BMI) < 30
* Ability to walk unaided for at least 10 minutes without major physical limitations

Exclusion Criteria:

* Presence of pain at the time of testing
* Self-reported diagnosed condition affecting mobility
* Known allergy to any component of the study cream
* Allergy to EMG electrode adhesives
* Inability to stand unassisted for more than 1 minute
* Inability to walk/run at the required speed and distance
* Weight exceeding 150 kg (due to treadmill limitations)
* Recent intake of:
* Analgesics (within 6 hours)
* Cigarettes (within 6 hours)
* Caffeine (within 2 hours)
* Skin lesions at the cream application site
* Pregnancy
* Failure to understand instructions
* Daytime pain reported by participant on day of experimentation

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Walk ratio | During intervention (pre/post cream application): for the mat, during a 2-minute free walk and for the treadmill, during a 5-minute treadmill walk with increases in speed every 30 seconds.
  Index that quantifies gait adaptations. Measured via GAITRite mat and Zebris treadmill.

SECONDARY OUTCOMES:
Gait Kinematics: Joint amplitudes | During intervention (pre/post cream application): for the mat, during a 2-minute free walk and for the treadmill, during a 5-minute treadmill walk with increases in speed every 30 seconds.
  High-resolution recordings of the walking tasks: sagittal plane of the lower limbs. Changes in the angles of the knee and ankle joints.
ECG/Heart Rate Variability (HRV) | During intervention (pre/post cream application): for the mat, during a 2-minute free walk and for the treadmill, during a 5-minute treadmill walk with increases in speed every 30 seconds.
  R-R interval variability during walking tasks.
Electrodermal Activity (EDA) | During intervention (pre/post cream application): for the mat, during a 2-minute free walk and for the treadmill, during a 5-minute treadmill walk with increases in speed every 30 seconds.
  Skin conductance during tasks.
Pain Catastrophizing (PCS) | Before intervention.
  Pain Catastrophizing Scale total score (0-52). Users rate 13 statements on a scale from 0 (not at all) to 4 (all the time).
Fear-Avoidance Beliefs (FACS) | Before intervention.
  Fear-Avoidance Components Scale total score (0-100). Users rate 20 statements from 5 (Strongly agree) to 0 (Strongly disagree).
Kinesiophobia (TSK) | Before intervention.
  Tampa Scale of Kinesiophobia total score (17-68). Users rate 17 statements in a scale from 1 (Strongly disagree) to 4 (Strongly agree).
Pain Severity (BPI) | Before intervention.
  The Brief Pain Inventory (Short Form) (BPI-SF) measures pain using three key scales: the Pain Severity Scale (ranging from 0 = "No pain" to 10 = "Pain as bad as you can imagine"), which assesses worst, least, average, and current pain over 24 hours; the Pain Interference Scale (0 = "Does not interfere" to 10 = "Completely interferes"), evaluating how pain affects daily activities like mood, work, and sleep; and the Pain Relief Scale (0% = "No relief" to 100% = "Complete relief"), indicating the effectiveness of pain treatments.
Self-Reported Pain (VAS) | 1 and 2. before and after application of the cream (intervention); 3. During the treadmill task: upon finishing the 1.3 m/s speed recording; 4. During the free-walking task: at half of the gait cycles; 5. Upon finishing all tasks.
  Visual Analog Scale (0-100 mm) for immediate pain intensity, where 0 = "No pain" and 100 = "Worst pain imaginable."
Gait Variability Index | During intervention (pre/post cream application): for the mat, during a 2-minute free walk and for the treadmill, during a 5-minute treadmill walk with increases in speed every 30 seconds.
  Step-to-step variability in stride time/length (coefficient of variation, %) derived from GAITRite/Zebris data.
Gait Symmetry Index | During intervention (pre/post cream application): for the mat, during a 2-minute free walk and for the treadmill, during a 5-minute treadmill walk with increases in speed every 30 seconds.
  Inter-limb asymmetry ratio (affected/unaffected side) for step length, stance time, and ground reaction forces (Zebris treadmill).

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Lelard, PhD, Study Director — Lecturer; Maryne Cozette, PhD, Study Director — Lecturer
Locations (1):
- Université de Picardie Jules Verne, Amiens, France

IPD SHARING:
Plan to Share IPD: No
Participants consented to data use only for this specific study under CERSTAPS-approved protocols.
  French and EU GDPR regulations prohibit broad sharing of pseudonymized sensor/video data that could potentially be re-identified (e.g., physical features in GoPro videos, unique gait patterns).

REFERENCES:
- [Background] Sarvestani M, Orakifar N, Mofateh R, Seyedtabib M, Karimi M, Mehravar M. The Association Between Lower Limb Joint Position Sense and Different Aspects of Gait Pattern in Individuals With Bilateral Knee Osteoarthritis. J Appl Biomech. 2025 Jan 3;41(2):107-116. doi: 10.1123/jab.2024-0207. Print 2025 Apr 1. PMID 39753124
- [Background] Bogen B, Moe-Nilssen R, Ranhoff AH, Aaslund MK. The walk ratio: Investigation of invariance across walking conditions and gender in community-dwelling older people. Gait Posture. 2018 Mar;61:479-482. doi: 10.1016/j.gaitpost.2018.02.019. Epub 2018 Feb 21. PMID 29494821
- [Background] Nishi Y, Osumi M, Sumitani M, Yozu A, Morioka S. Kinematic changes in goal-directed movements in a fear-conditioning paradigm. Sci Rep. 2021 May 27;11(1):11162. doi: 10.1038/s41598-021-90518-7. PMID 34045515
- [Background] Karos K, Meulders A, Gatzounis R, Seelen HAM, Geers RPG, Vlaeyen JWS. Fear of pain changes movement: Motor behaviour following the acquisition of pain-related fear. Eur J Pain. 2017 Sep;21(8):1432-1442. doi: 10.1002/ejp.1044. Epub 2017 Apr 25. PMID 28444803
- [Background] Horvath A, Koteles F, Szabo A. Nocebo effects on motor performance: A systematic literature review. Scand J Psychol. 2021 Oct;62(5):665-674. doi: 10.1111/sjop.12753. Epub 2021 Jun 18. PMID 34145580